CLINICAL TRIAL: NCT07342777
Title: EXpain - Is Exercise an Effective Non-pharmacological Analgesic Treatment in People With Multiple Sclerosis?
Brief Title: EXpain Trial - Exercise an a Non-pharmacological Pain-relieving Treatment in People With Multiple Sclerosis
Acronym: EXpain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EXpain Trial
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-08

CONDITIONS: Multiple Sclerosis; Chronic Pain; Neuropathic Pain
Keywords: Exercise therapy; multiple sclerosis; pain; chronic pain; neuropathic pain; non-pharmacological analgesics; resistance exercise; physical exercise; Rehabilitation; Mixed type pain
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain; Neuralgia; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: See study description for details
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercise group (Experimental): Participants must have chronic pain (NRS ≥ 3) when enrolled and furthermore meet eligibility criteria.
  Intervention: 12 weeks of progressive resistance exercise followed by 12 weeks of usual care
  Interventions: Other: Progressive resistance exercise
- Waitlist group (Experimental): Participants must have chronic pain (NRS ≥ 3) when enrolled and furthermore meet additional eligibility criteria. Intervention: 24 weeks of usual care followed by 12 weeks of progressive resistance exercise.
  Interventions: Other: Usual Care followed by progressive resistance exercise

INTERVENTIONS:
Other: Progressive resistance exercise — Participants assigned to this arm will undergo 12 weeks of progressive heavy-load resistance exercise, with 5 sessions over a 2-week period (equaling a total of 30 sessions). Each session will commence with a 5-minute warm-up using a bicycle ergometer. The training program will consist of machine-based exercises, including leg press, knee extensions, hamstring curls, seated calf raises, chest press, and lateral pull-down. Progression will be ensured through an increase in the number of sets (from 3 to 4, interspersed by 1-2 minutes of rest) for each exercise along with an increment in intensity (from 15 Repetition Maximum (RM) towards 8RM.
  Arms: Resistance exercise group
Other: Usual Care followed by progressive resistance exercise — Participants assigned to this arm will undergo 24 weeks of waitlist control. The control group will continue their habitual lifestyle and usual care throughout the whole period. After 24 weeks, the waitlist control group will undergo the same progressive resistance exercise regimen as described in the intervention group.
  Arms: Waitlist group

SUMMARY:
The primary goal of this study is to test whether 12 weeks of progressive resistance exercise is an effective non-pharmacological treatment for reducing pain in people with multiple sclerosis and chronic pain.

The study will be a randomized controlled trial with multiple training sites. After baseline testing, participants will be randomly assigned to either a 12-week progressive resistance exercise intervention followed by a 12-week follow-up period or to a 24-week waitlist control group that receives usual care.

It is hypothesized that people with multiple sclerosis and chronic pain who receive the intervention will experience greater reductions in pain (i.e., clinically relevant reductions) compared to the waitlist control group (primary hypothesis), and that this pain reduction will be preserved after a 12-week follow-up period (secondary hypothesis).

DETAILED DESCRIPTION:
Purpose and Hypotheses:

The main purpose of this project is to understand the impact of pain in people with multiple sclerosis, how exercise may affect pain symptoms, and whether these effects depend on the underlying pain mechanisms and/or biopsychosocial factors.

The purpose of the main study (study 2) is to test the hypotheses that:

People with MS receiving 12 weeks of resistance exercise will experience superior average analgesic effects (i.e., clinically relevant reductions), compared with MS controls receiving usual care (primary hypothesis), and this analgesic effect will be preserved after a 12-week follow-up period (secondary hypothesis).

The purpose of studies 1,3, 4, and 5 is to test the hypotheses that:

* In people with MS, pain severity will be negatively associated with physical activity, everyday life, walking ability, sleep quality, and/or quality of life, while being positively associated with anxiety, depression, and/or fatigue (study 1).
* People with MS suffering from mixed type pain will experience greater analgesic effects after 12 weeks of resistance exercise compared to people with MS suffering from neuropathic pain (study 3).
* A single bout of resistance and aerobic exercise will acutely induce an analgesic effect as well as a reduction in pain sensitivity immediately after an exercise session, compared with pre-exercise levels, transiently disappearing over the next 15 minutes (study 4).
* Our multifactorial model, incorporating biomarkers, sensory profiles, pain phenotypes, and patient-reported outcomes, is hypothesized to explain the variability of the analgesic effects of resistance exercise to a large extent (i.e., approximately 81%1)(study 5).

Background:

Multiple sclerosis (MS) is a chronic neurodegenerative demyelinating disorder of the central nervous system with profound physical, cognitive, and social consequences. Symptomatic treatment to address these consequences and to improve the quality of life in people with multiple sclerosis (pwMS) is thus essential. One symptom that significantly affects the quality of life in pwMS is pain. Pain is one of the most common symptoms in MS and has recently been estimated to affect as many as 75% of all pwMS. The International Association for the Study of Pain (IASP) has proposed three mechanistic descriptors that may identify different primary pain types or mechanisms, which may exist alone or in combination (i.e., mixed-type pain): 1) Neuropathic pain, defined as pain caused by lesions or disease of the somatosensory nervous system 2) Nociceptive pain, defined as an appropriate pain arising from the activation of nociceptors in non-neural tissue. 3) Nociplastic pain, defined as the presence of pain despite any apparent damage to neuronal or non-neuronal tissue. It is not possible to exclude neuropathic pain in MS, considering the neurodegenerative nature of the disease. However, it may not be the only/or dominant descriptor underlying the experienced pain. Thus, pain will henceforth be referred to as either neuropathic or mixed in the current project.

The majority of current analgesic (pain relieving) treatments include pharmacology and account for approximately 30% of the total medication in MS 7. Pain medication is known to be costly and has extensive adverse effects. Thus, cost-effective non-pharmacological analgesic treatment options without substantial side effects are highly warranted in MS.

Exercise might be exactly such an option. In the general population, exercise has been shown to improve pain symptoms, be cost-effective, and present few, if any, adverse effects beyond exercise-induced soreness. Exercise has been observed to have both acute and chronic beneficial effects on perceived pain in other populations. In neurodegenerative populations, only limited evidence exists, but analgesic effects of exercise have been reported in Parkinson's Disease. A systematic review in 2019 identified 10 exercise studies that had pain as an outcome, which overall suggested a chronic analgesic effect of exercise In MS. However, across these 10 exercise studies, pain was assessed as a secondary outcome, and participants were not recruited based on their initial baseline pain status (i.e., some participants did not experience pain symptoms at study entry).

An important distinction relates to the potential different acute and chronic analgesic effects obtained following different exercise modalities. In other populations, evidence points to resistance exercise as one of the most potent modalities in terms of achieving analgesic effects, although verifying studies in MS are lacking. Examining the efficacy of basic exercise modalities, such as resistance exercise, while further elucidating underlying mechanisms, appears highly relevant in order to improve pain management in people with MS.

In the majority of treatments, a response heterogeneity has been observed, and this also seems to be the case for analgesic treatments. Studies based on surgical and pharmacological treatments of pain have had success identifying that different pain biomarkers, such as inflammatory biomarkers, sensory profiles, and patient-reported outcomes, can predict the analgesic effects in patients. Additionally, we have seen that combining different pain biomarkers yields a larger predictive value than only assessing a single pain biomarker with a study showing such models to explain up to 81% of the variability of clinical pain intesity. However, such predictive models have not yet been adopted in any exercise treatments. Exploring how analgesic effects induced by resistance exercise are associated with - or can even be predicted by - relevant factors appears highly relevant to facilitate and prescribe personalized pain treatment.

In summary, research investigating whether exercise holds the potential to induce analgesic effects in people with MS affected by pain, both in the long-term (i.e., the pain level after a period of regular exercise sessions) and/or acutely (i.e., effects observed immediately after a single exercise session), is highly warranted. Furthermore, insights into underlying characteristics and how they affect the analgesic potential of resistance exercise are necessary to optimize personalized treatment prescription in MS.

Methods:

Study Design To expand our current understanding of the effects of exercise on pain in MS, we have designed a assessor blinded randomized controlled trial (RCT) with follow-up (study 2) with four integrated sub-studies: an initial cross-sectional study (study 1), an exploratory interventional study (study 3) an acute interventional study (study 4) and yet an exploratory interventional study (study 5) (see figure Patient and public involvement

Study 1: This is a cross-sectional survey-based study (i.e., relying on self-reporting) using Redcap, investigating the association between pain severity (NRS0-10 ≥3 ) and physical activity, walking ability, sleep quality, anxiety and depression, fatigue, as well as quality of life. This includes a comparison between people with MS having severe pain (NRS0-10 ≥3) and having no (NRS0-10 = 0) mild pain (NRS0-10 <3). Furthermore, this study will serve as a screening tool for study 2.

Study 2: ("the main study"): Upon interest and fulfillment of eligibility criteria, potential participants identified via study 1 with pain levels NRS0-10 ≥3 will be enrolled and randomized to either 12 weeks of progressive resistance exercise, succeeded by a 12-week follow-up period, or to a 24-week waitlist control group. During the follow-up period, participants will be encouraged to continue exercising independently and will be asked to keep an exercise diary. The control group will proceed with their habitual lifestyle during the 24 weeks.

Study 3: Participants from the waitlist control group in study 2 will, after 24 weeks, be enrolled into the same 12-week intervention as provided in study 2. The control group data derived from weeks 24 to 36 will be pooled with data from the intervention group in study 2, enabling an exploratory analysis of potential phenotype-dependent differences in the analgesic effect of exercise on pain. This design will furthermore ensure that all participants are enrolled in an exercise intervention (either from weeks 0-12 or 24-36), which is likely to promote study adherence.

Study 4: To determine the acute effects of exercise on pain, data on pressure pain threshold (PPT) and pain severity (NRS0-10) will be extracted immediately before and after a bout of resistance exercise during studies 2 and 3. Furthermore, pain severity will be monitored at 5-, 10-, and 30-minute post-exercise. To investigate any potential modality-dependent variations in the acute effects of exercise on pain, the described protocol will be further applied to a 45-minute bout of aerobic exercise. Moreover, measurements of PPT and pain severity will be applied to a bout of isometric exercise at baseline, post-assessment, and at follow-up to assess potential changes in the acute pain response to exercise following 12 weeks of resistance exercise.

Study 5: To evaluate the predictive value of a multi-factorial approach on the effect of exercise on pain, blood samples, sensory profiles, and patient-reported outcome measures (PROMs) will be collected at baseline and after interventions in both groups (i.e., T0 + T12 for the intervention group and T24 + T36 for the wait-list group).

Interventions:

All of the following interventions will be supervised and tailored to the individual participant´s absolute strength, ensuring equal relative intensity throughout the project.

Main intervention - Progressive resistance exercise (Chronic effect) Description and progression Load (RM): 15 (week 1-3), 12 (week 4-6), 10 (week 7-9), 8 (week 10-12) Number of repetitions: 12 (week 1-3), 10-12 (week 4-6), 8-10 (week 7-9), 6-8 (week 10-12) Number of sets: 3 (week 1-6), 4 (week 7-12) Contraction type: Isotonic (concentric and eccentric) Recovery time between sessions (hours): >48

Progressive resistance exercise (Acute effect) At session 2 during week 1, participants will undergo the aforementioned resistance exercise regimen consisting of 12 repetitions of 15 RM for 3 sets, interspersed by 2-3 minutes.

Aerobic exercise (Acute effect) At training session 4 during week 2, participants will undergo a separate bout of aerobic exercise consisting of 30 minutes at 75% - 80% of estimated HRmax, using a bicycle ergometer. The session will commence with a 5-minute warm-up and terminate with a 5-minute cool-down using the same bicycle ergometer.

Isometric Exercise (Acute effect) To determine the acute pain response to exercise and assess potential changes following 12 weeks of resistance exercise, participants will undergo a single bout of isometric exercise of the lower extremities using a leg press dynamometer at an intensity of 30% of maximal voluntary contraction for 90 seconds at baseline and post-intervention (T0+T12 or T24+T36).

Outcomes:

See section "Outcome Measures" for specifications. Additionally, contact information, demographic information, health and medication information as well as blood samples will be obtained.

Statistical considerations:

To assess differences between participants experiencing moderate to severe pain and participants experiencing mild to no pain with regard to selected parameters, a linear mixed model will be applied in study 1. To analyse the effects of exercise on pain severity (chronic and acute), and potential phenotype-dependent differences, a linear mixed-effects intention-to-treat model (including all participants enrolled at baseline) will be applied to study 2, 3, and 4. Finally, to describe the chronic postinterventional pain severity in study 5, a supervised multivariate data analysis with "Data Integration Analysis for Biomarker Discovery" using Latent Components (DIABLO) will be applied.

The main study (study 2) will be powered based on the primary outcome measure NRS0-10, relying on data from previous exercise studies in MS and other relevant populations24,52-54. A two-sample two-sided power calculation resulted in a total of n=58 subjects, which will be expected to be enrolled in each group (α=0.05; power=0.9; control pre-post change 0.3 NRS0-10 score and SD=1.8; exercise pre-post change 1.2 NRS0-10 score and SD=1.8; dropout rate=15%). Hence, a total of 116 participants will be enrolled in the present study.

Randomization:

After baseline assessment of participants, they will be randomized to either the intervention or waitlist control group using a 1:1 ratio. A computer-generated list of random numbers will be conducted in the Research Electronic Data Capture (REDCap) system. The randomization will be stratified by site and will be blinded to outcome assessors.

Perspectives:

The findings of this project have the potential to establish progressive resistance exercise as an effective, safe, and accessible treatment of pain in people with MS and elucidate how this effect may be distinct depending on pain phenotype, inflammatory biomarkers, as well as psychological and physical states. Furthermore, it will examine the acute effects of resistance and aerobic exercise on pain, thereby advancing the understanding of their interrelationship in this population. Finally, insights into the impact of pain in MS will highlight key considerations for pain management. Conclusively, this study has the potential to transform pain management for people with MS suffering from pain worldwide by reducing reliance on pharmacological analgesics and, as a result, minimizing associated adverse effects and lowering societal costs.

ELIGIBILITY:
Inclusion criteria: Average pain levels of >3 on the Numerical Rating Scale from 0-10 (NRS0-10), age ≥ 18 years, a valid MS diagnosis (ICD-10 code: G35), ability to self-transport to test and exercise.

Exclusion Criteria: Pregnancy, Diabetes, neurological or other comorbidities that hinder participation in the study, relapse within the past 2 months, classified as high cardiovascular risk according to the American College of Sports Medicine´s guidelines, and participation in structured exercise over the past 3 months (≥ 2 sessions/week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in pain severity | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  Subjective average pain severity over the past 7 days measured using a Numerical Rating Scale from 0 to 10 (NRS0-10)

SECONDARY OUTCOMES:
Change in Brief Pain Inventory (BPI) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Brief Pain Inventory assesses pain severity and its impact on daily life, encompassing pain intensity, interference with activities, mood, and sleep. Additionally, it inquires about pain distribution and management strategies. Scores are calculated based on responses, with higher scores indicating more severe pain and greater interference with daily activities
Change in Graded Chronic Pain Scale (GCPS-R) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Graded Chronic Pain Scale (GCPS-R) assesses chronicity of pain (i.e., persisting pain for at least 3 months) and its severity through two overall dimensions: pain intensity and pain-related disability in the past 7 days. Moreover, it grades the severity of chronic pain from 0 (no pain) to 4 (high disability severely limiting).
Change in Douleur Neuropathique 4 questions (DN4) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Douleur Neuropathique 4 Questions (DN4) is a simple screening tool for possible indications of neuropathic pain (note: it does not provide a diagnosis). It consists of 7 self-reported items and a clinical examination consisting of three items. Scores ≥ 4/10 indicate neuropathic pain. DN4 will be included, but will not stand alone, in the diagnosis of neuropathic pain in participants.
Change in physical activity (Baecke Habitual Physical Activity Questionnaire) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Baecke Habitual Physical Activity Questionnaire is a tool used to assess an individual's level of physical activity in their daily life. It consists of a series of questions covering three domains: work-related physical activity, sports-related physical activity, and leisure-time physical activity. Each domain assesses the frequency, intensity, and duration of physical activities performed by the individual. The questionnaire aims to capture the overall level of physical activity and its distribution across different life domains. Higher scores indicate a higher level of physical activity.
Change in Hospital Anxiety and Depression Scale (HADS) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Hospital Anxiety and Depression Scale (HADS) consists of 14 items, divided evenly between anxiety (7 items) and depression (7 items), with each subscale scored from 0 to 21. Scores of 8-10 suggest a moderate level of symptoms, while scores above 11 indicate a substantial symptom burden that likely corresponds to a clinical diagnosis
Change in Pittsburgh Sleep Quality Index (PSQI) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Pittsburgh Sleep Quality Index is a questionnaire used to assess sleep quality over a one-month time interval. It comprises 19 items covering seven components: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored on a scale from 0 to 3, with higher scores indicating poorer sleep quality. The total score ranges from 0 to 21.
Change in Multiple Sclerosis Walking Scale-12 (MSWS-12) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The 12-Item Multiple Sclerosis Walking Scale (12-MSWS) is a validated questionnaire designed to capture the impact of multiple sclerosis on walking ability. It evaluates how the condition affects walking and balance during daily activities, such as climbing stairs, walking speed, and dependence on walking aids, over the past two weeks. Each item is rated on a five-point Likert scale (1 = not at all to 5 = extremely), and responses are converted into a percentage score, with higher scores indicating a greater impact
Change in Modified Fatigue Impact Scale (MFIS) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Modified Fatigue Impact Scale (MFIS) is a self-report questionnaire designed to assess the perceived impact of fatigue. It evaluates how fatigue has affected physical, cognitive, and psychosocial functioning over the past four weeks. The MFIS consists of 21 items rated on a Likert scale, with higher scores indicating greater fatigue-related impact. Subscale scores can be calculated for physical, cognitive, and psychosocial domains, and combined to produce a total score ranging from 0 to 84, with higher scores indicating greater impact.
Change in MS-impact Scale-12 (MSIS-29) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Multiple Sclerosis Impact Scale (MSIS-29) is a 29-item self-report questionnaire designed to measure MS-related quality of life via the physical and psychological impact of multiple sclerosis on daily life over the preceding two weeks. It comprises two subscales: a physical impact scale (20 items) and a psychological impact scale (9 items). Each item is rated on a five-point scale (1 = not at all to 5 = extremely). Subscale scores are calculated by summing item responses and transforming them into a 0-100 scale, with higher scores indicating greater disease impact and poorer health status. The MSIS-29 is widely used in both clinical practice and research as a patient-reported outcome measure
Change in daily fluctuations in pain severity | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  To detect potential fluctuations in pain, participants will rate themselves (NRS0-10) every 2 waking hours for 3 consecutive days following every test session using automated texts.
Change in daily fluctuations in fatigue severity | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  To detect potential fluctuations in fatigue, participants will rate themselves (NRS0-10) every 2 waking hours for 3 consecutive days following every test session using automated texts.
Change in Clinical Sensory Test (CST) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  To assess the sensory profile of participants, a Clinical Sensory Test (CST) battery will be conducted, containing thermal stimuli using a metal object at temperatures of 38-42°C and cold 17-21°C in addition to mechanical stimuli using light touch (cotton/sensobrush), pinprick (toothpick), and vibration (tuning fork 128 Hz). To determine sensory abnormalities, all stimuli will be applied to a non-painful site as well as a painful site, allowing for a comparison of perception between the two. CST will be included, but will not stand alone, in the diagnosis of neuropathic pain in participants.
Change in pressure Pain Detection Threshold and pressure Pain Tolerance Threshold | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  To assess participant´s pressure pain sensibility, pressure Pain Detection Threshold (PDT) and pressure Pain Tolerance Threshold is measured using cuff pressure algometry. A pressure cuff is strapped around the lower leg of participants and the pressure is increased gradually at a rate of 1 kPa/s. The subject will be instructed to rate the pain intensity continuously a the electronic Visual Analog Scale (VAS) until the tolerance level is reached. Further, the subject is instructed to press a stop button when the tolerance level is reached, which will release the pressure immediately. The pressure pain threshold (PDT) is defined as the pressure at which the VAS score exceeds 1 cm, and the pressure pain tolerance threshold (PTT) is defined as the pressure at which the participant presses the stop button.
Change in Temporal Summation of Pain (TSP) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  Temporal Summation of Pain (TSP) reflects the facilitatory capabilities of the nociceptive system. It will be investigated using cuff pressure algometry. A total of 10 repeated mechanical pressure stimuli will be delivered at 0.5 Hz (1-s stimulus duration and 1-s interstimulus intervals) to the test limb. During the 10 repeated stimuli, the subjects will continuously rate the pain intensity on the electronic VAS.
Change in Conditioned Pain Modulation (CPM) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  Conditioned Pain Modulation reflects the inhibitory capabilities of the nociceptive system. CPM will be measured in succession of the PDT, PTT and TSP measurements. An additional tourniquet cuff is fitted around the contralateral limb and applies a painful tonic stimulus (conditioning stimulus). Simultaneously, the other cuff applies a gradually increasing pressure of 1kPa/s (test stimulus), as described in PDT and PTT. Both the conditioning and test stimuli will be terminated when the subject presses the stop button. CPM will be defined as the difference between the stimulus during and before the conditioned pain (i.e., "during" minus "before").
Change in Exercise Induced Hypoalgesia (EIH) and EIH-respons associated with a realistic bout of resistance exercise (aprox. 45 min full body workout) as well as a realistic bout of aerobic exercise on a bicycle ergometer (45 min at 70% of HRmax). | Intervention group: Baseline, 12 week post test, 24 weeks follow-up Waitlist group: Baseline, 12 weeks post test, 24 weeks follow-up/baseline, 36 weeks post test.
  Exercise induced Hypoalgesia (EIH) is a phenomenon that is defined as a reduction in pain pressure threshold after a bout of exercise. To measure this acute effect of exercise, a 1 cm² flat probe is placed perpendicular to the skin locally (i.e., exercising limb) at the middle of the dominant quadriceps muscle (15 cm proximal to the base of patella) and remotely (i.e., non-exercising limb) at the upper trapezius of the non-dominant side. If pain is present in the dominant leg or trapezius of the non-dominant side, data will be collected from the opposite limb to avoid potential disturbance. Hereafter, an increasing pressure of 30 kPa/s is applied until the participant perceives the pressure as painful and ceases the test by pressing a button. This point is defined as Pressure Pain Threshold (PPT). This process is repeated thrice at each site, and the average PPT will be used for further analysis before an after exercise. Furthermore, pain severity will be measured using the NRS0-10.
Change in muscle strength of the lower extremities | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  A custom-built leg press dynamometer will be used to measure muscle strength through maximal voluntary contractions. The patient will continue until a maximum has been found. Appropriate breaks are held between the repetitions.
Change in Six Minute Walk Test (6MWT) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The Six Minute Walk Test (6MWT) is a simple and widely used measure of functional exercise capacity. After the six minutes have elapsed, the total distance walked by the participant is recorded in meters. Longer distances indicate better functional exercise capacity and endurance.
Change in 9-Step Stair Ascend (9SSA) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  The 9-Step Stair Ascend (9SSA) measures functional capacity an is furthermore an indirect measure of power.
Changes in 5-times Sit-To-Stand (5STS) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  5-times Sit-To-Stand (5STS) is a measure of physical function and correlates well with in daily life. During this test the participant are instructed to get up from a chair and sit back down five times as quickly as possible.
Changes in physical activity (Accelerometery) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  Accelerometery objectively measures the level of physical activity. An accelerometer will be placed on the outside of the participants upper thigh as this placement has proven more accurate. It is to be worn for 7 consecutive days following each test-session.
Changes in C-reactive Protein (CRP) | Intervention group: Baseline, 12 weeks post test Waitlist group: Baseline, 36 weeks post test.
  The study will investigate inflammatory factors using plasma samples collected from the participants. The analysis will consist of two main steps: analysis of C-Reactive Protein (CRP) through ELISA, and analysis of 96 Inflammatory Markers with the OLINK Inflammatory Panel. ELISA stands for Enzyme-Linked Immunosorbent Assay. It is a laboratory technique used to detect and quantify specific proteins, like antibodies or antigens, in a sample. The assay uses a solid-phase type of enzyme immunoassay (EIA) to detect the presence of a ligand (commonly a protein) in a liquid sample using antibodies directed against the protein to be measured. The present technique has been used largely in the past years and represents a gold standard for diagnostics.
Changes in inflammatory biomakers | Intervention group: Baseline, 12 weeks post test Waitlist group: Baseline, 36 weeks post test.
  Analysis of 96 Inflammatory Markers with OLINK Inflammatory Panel will be performed. The OLINK panel is an assay that uses proximity extension assay (PEA) technology. In this method, pairs of antibodies linked to DNA probes are used to quantify specific proteins. When the antibodies bind to their target proteins, the DNA probes come into proximity and generate a quantifiable signal.
Changes in microRNA´s (miRNA's) | Intervention group: Baseline, 12 weeks post test Waitlist group: Baseline, 36 weeks post test.
  MicroRNA´s has been suggested to have inflammatory properties and to be positively correlated with pain. The evaluation of circulating miRNAs will follow a two-phase approach: a discovery phase using Next-Generation Sequencing (NGS) and a validation phase using quantitative real-time PCR (qPCR).
Change in pain distribution (Navigate Pain) | Intervention group: Baseline, 12 weeks post test, 24 weeks follow up test. Waitlist group: Baseline, 12 weeks post test, 24 weeks follow up/ baseline test, 36 weeks post test.
  Navigate Pain is a digital pain distribution map where participants can engrave the exact areas where they are experiencing pain. Moreover, it enables the participants to further characterize their pain using relevant descriptors corresponding to the engraved areas.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Prior to analysis, pseudonymized whole blood and plasma samples will be shipped by project personnel to Aalborg University, Selma Lagerløfs Vej 249 and stored in a locked -70°C freezer until they are analyzed, ensuring sample integrity and minimizing technical bias. miRNA analysis will be carried out by QIAGEN Genome Service, located in Hilden, Germany. For this purpose, 200/400 ul per sample, completely anonymized, will be shipped in cryo boxes from Aalborg University to QIAGEN in Hilden, Germany.
  Analysis of 96 Inflammatory biomarkers will be performed by BioXpedia A/S, Palle Juul-Jensens Blvd. 82, 8200 Aarhus N, or carried out by Associate Professor Rocco Giordano at Aalborg University, SUND, Selma Lagerløfs Vej 249. All of the abovementioned analyses will be run following and respecting GDPR related laws.
  Data on pain distribution will be shared with Navigate Pain (Aglance Solutions) and stored on Europe-based servers complying with GDPR.
Supporting Information: Study Protocol, ICF
Time Frame: Sharing of data will commence February 2026 and is expected to terminate within a 5-year period following August 2028.
Access Criteria: Data will be accessible exclusively to authorized personnel on encrypted servers. Data collection and data management will be conducted solely by trained staff operating under restricted access privileges.

REFERENCES:
- [Background] Rosner J, de Andrade DC, Davis KD, Gustin SM, Kramer JLK, Seal RP, Finnerup NB. Central neuropathic pain. Nat Rev Dis Primers. 2023 Dec 21;9(1):73. doi: 10.1038/s41572-023-00484-9. PMID 38129427
- [Background] Heesen C, Bohm J, Reich C, Kasper J, Goebel M, Gold SM. Patient perception of bodily functions in multiple sclerosis: gait and visual function are the most valuable. Mult Scler. 2008 Aug;14(7):988-91. doi: 10.1177/1352458508088916. Epub 2008 May 27. PMID 18505775
- [Background] Vaegter HB, Jones MD. Exercise-induced hypoalgesia after acute and regular exercise: experimental and clinical manifestations and possible mechanisms in individuals with and without pain. Pain Rep. 2020 Sep 23;5(5):e823. doi: 10.1097/PR9.0000000000000823. eCollection 2020 Sep-Oct. PMID 33062901
- [Background] Demaneuf T, Aitken Z, Karahalios A, Leong TI, De Livera AM, Jelinek GA, Weiland TJ, Marck CH. Effectiveness of Exercise Interventions for Pain Reduction in People With Multiple Sclerosis: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Arch Phys Med Rehabil. 2019 Jan;100(1):128-139. doi: 10.1016/j.apmr.2018.08.178. Epub 2018 Sep 19. PMID 30240593
- [Background] Yamout B, Issa Z, Herlopian A, El Bejjani M, Khalifa A, Ghadieh AS, Habib RH. Predictors of quality of life among multiple sclerosis patients: a comprehensive analysis. Eur J Neurol. 2013 May;20(5):756-64. doi: 10.1111/ene.12046. Epub 2013 Jan 8. PMID 23294397
- [Background] Giordano R, Arendt-Nielsen L, Gerra MC, Kappel A, Ostergaard SE, Capriotti C, Dallabona C, Petersen KK. Pain mechanistic networks: the development using supervised multivariate data analysis and implications for chronic pain. Pain. 2025 Apr 1;166(4):847-857. doi: 10.1097/j.pain.0000000000003410. Epub 2024 Sep 18. PMID 39297729